CLINICAL TRIAL: NCT07286955
Title: SAFEGUARD: Life Skills Training for Soldiers Arriving at Their First Duty Location
Brief Title: Life Skills Training for Soldiers Arriving at Their First Duty Location
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Defense Health Agency (U.S. Federal Agency); Harvard University (Other); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USUHS.2025-162; Federal Award # HU00012520025 (Other Grant/Funding Number: Assistant Secretary of War for Health Affairs)
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Risk Reduction Behavior; Suicide Prevention; Risky Behavior; Mental Health; Resilience; Performance at Work
Keywords: Military Health; Suicide Prevention; Harmful Behaviors; Life Skills Training; First Duty Location; Active-duty Military; Risk Reduction; Prevention; Level Up
MeSH Terms: conditions — Risk Reduction Behavior; Suicide Prevention; Psychological Well-Being | interventions — engage 8200

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Level Up Program (Experimental): The Level Up program is a hybrid intervention combining interactive learning, mobile/online technology, personalized coaching, and on-demand virtual booster sessions. The evidence-based training program was designed to build life skills and coping strategies that can protect against suicide, other harmful behaviors, poor work performance, and premature separation during a Soldier's first duty assignment.
  Interventions: Behavioral: Level Up
- ENGAGE Training (Active Comparator): ENGAGE is an existing single session Army bystander intervention program. The training program is based on bystander intervention and prosocial behavior research.
  Interventions: Behavioral: ENGAGE

INTERVENTIONS:
Behavioral: Level Up — The Level Up program components include:
  * A 90-minute live group session during Soldiers' in-processing week at their first duty station
  * A mobile app/online platform/workbook with brief, interactive self-guided exercises in core skill areas (e.g., managing stress, tactical thinking, healthy relationships)
  * Personalized coaching via messages from trained Level Up staff during the first month of app use
  * Virtual booster sessions over one year, focused on practical domains like finances, leadership, promotion tips, and personal relationships
  Other Names: Life Skills
  Arms: Level Up Program
Behavioral: ENGAGE — ENGAGE training is a single 90-minute workshop aimed at developing leadership skills and confidence in handling professional and personal confrontations.
  Arms: ENGAGE Training

SUMMARY:
This project will evaluate the effectiveness of Level Up: Boost Your Life Skills ("Level Up"), a strengths based, military-specific life skills training program. The goal is to determine whether Level Up can decrease suicidal-related behaviors (SRBs) and other harmful behaviors, improve mental health, enhance job performance, and reduce early military separation. The Level Up program components will be made available to participants through an online platform or mobile app that can be downloaded onto their personal mobile devices. These training materials will help Soldiers learn and practice skills. The Level Up program will also involve personalized messages from a Level Up trainer and virtual booster sessions. Soldiers arriving at their first duty location will be randomized to receive either Level Up or a single session Army bystander intervention program. Participants will complete baseline and follow up surveys 1, 3, and 6 months post-baseline.

DETAILED DESCRIPTION:
Suicide remains a leading cause of death among Soldiers, especially those 17-24 years old in their first year of military service. This time is also marked by high rates of other harmful behaviors and of early separation from the Army. The Army invests billions of dollars in recruiting and training, yet many new Soldiers leave the service early or experience serious events like suicidal behaviors. Exposure to situational stressors involving such areas of life as romantic relationships and finances increases risk for suicide and other harmful behaviors. Implementing universal training programs to prevent these types of negative outcomes before they arise have enormous potential to bolster the mental toughness of new Soldiers during this difficult transition. The proposed project aims to prevent suicide-related behaviors (SRBs) and other behaviors qualifying for a Serious Incident Report (SIR) through an innovative, universal life skills program delivered at a critical transition point in Soldiers' careers-their first duty assignment. By focusing on this particularly high-risk period, this project seeks to reduce SRBs and related harmful behaviors among U.S. Army Soldiers. The proposed project will test the effectiveness of a recently developed, evidence-based training program designed to build life skills and coping strategies that can protect against suicide, other harmful behaviors, poor work performance, and premature separation during a Soldier's first duty assignment.

This project will evaluate the effectiveness of Level Up, a strengths based, military-specific life skills training program. The goal is to determine whether Level Up can decrease suicidal thoughts and behaviors, improve mental health, enhance job performance, and reduce early military separation. Previous studies show that building skills like stress management, problem-solving, and healthy communication can protect against SRBs and related problem behaviors. However, many of these programs failed to show long-term impact, partly due to limited engagement. Level Up is designed to overcome these limitations by combining interactive learning, mobile technology, personalized coaching, and on-demand virtual booster sessions. This hybrid format is intended to help Soldiers refresh their skills and engage with content at their preferred pace and rhythm. The Level Up program components include: 1) a 90-minute live group session during Soldiers' in-processing week at their first duty station, 2) a mobile app/online platform/workbook with brief, interactive self-guided exercises in core skill areas (e.g., managing stress, tactical thinking, healthy relationships), 3) personalized coaching via messages from trained staff during the first month of app use, and 4) virtual booster sessions over one year, focused on practical domains like finances, leadership, promotion tips, and personal relationships. Soldiers will be randomized to receive either Level Up or Engage, an existing single session Army bystander intervention program that will serve as a comparison training.

The Level Up program content draws from evidence-based psychological methods such as Cognitive Behavioral Therapy, Acceptance and Commitment Therapy, and motivational coaching adapted to fit military culture and tailored to be relevant, accessible, and engaging for newly assigned junior-ranking Soldiers, a group at high risk for suicide and other serious behavioral issues. By equipping them with essential life skills and support during their first year of service, the program aims to reduce SRBs and other behaviors qualifying for SIRs, develop psychosocial skills, and increase career success and satisfaction.

If effective, Level Up could be implemented Army-wide as a universal prevention program to improve mental health, readiness, and retention. There are minimal risks as the interventions are educational, although some participants may experience brief emotional discomfort during skill practice or reflection. All participants can opt out at any time, and all are provided with resources and additional support as needed. This study could have a transformative impact on military suicide prevention efforts, especially during early service when Soldiers are most vulnerable. By evaluating this scalable program in a large, real-world setting, the research will provide clear evidence about its benefits for reducing suicide and improving readiness. Results will also support development of predictive tools to identify which Soldiers may benefit most from added support. Findings will be shared across the Department of Defense to inform policy, training, and future resilience-building programs-ultimately improving the health, performance, and quality of life of Soldiers across the Force.

ELIGIBILITY:
Inclusion Criteria:

* Active duty Soldiers arriving at a military installation located in the South Central U.S. for their first duty location who are attending reception center activities

Exclusion Criteria:

* Soldiers who are not available to attend the in-person training
* Soldiers who are under the age of 18 years old
* Soldiers who do not have a smart phone that supports installation of the mobile app

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of any harmful behavior | Within the 12 months after intervention randomization
  The occurrence of any harmful behavior, either self-reported in follow up surveys or administratively reported
The occurrence of any suicide-related behavior | Within the 12 months after intervention randomization
  The occurrence of any suicide-related behavior, either self-reported in follow up surveys or administratively reported

SECONDARY OUTCOMES:
The occurrence of any premature separations from service | Within the 12 months after intervention randomization
Poor performance as indicated either by written reprimands, designations in the NCOER, a corrective action plan, remedial training, flagging actions, demotion, Article 15, or barred reenlistment | Within the 12 months after intervention randomization
Personal deployment readiness | Within the 6 months after intervention randomization
  Walter Reed Army Institute of Research Land Combat Survey; Scale ranges from 4-20; Higher scores indicate higher perceived readiness
Emotionality | Within the 6 months after intervention randomization
  Emotion Reactivity Scale (ERS) ; Scale ranges from0-4; Higher scores indicate higher of each maladaptive trait
Job satisfaction | Within the 6 months after intervention randomization
  3-item Job Satisfaction Scale; Scale ranges from 3-15; Higher scores indicate higher perceived job satisfaction
Depression symptom severity | Within the 6 months after intervention randomization
  Patient Health Questionnaire-2 (PHQ-2); Scale ranges from 0-8; Higher scores indicate more severe symptoms
Anxiety symptom severity | Within the 6 months after intervention randomization
  Generalized Anxiety Disorder-2 (GAD-2); Scale ranges from 0-8; Higher scores indicate more severe symptoms
Incidence of traumatic brain injuries | Within the 6 months after intervention randomization
  Number of traumatic brain injuries; based on the Army STARRS Surveys; No scale range; number indicates greater number of traumatic brain injuries
Lifetime history of various mental/emotional health problems | Within the 6 months after intervention randomization
  Family History Screen (FHS); Scale ranges from 0-1; 0=No; 1=Yes
Chronic stress severity | Within the 6 months after intervention randomization
  Personal Life Stress Scale (PLS); Scale ranges from 0-50; Higher scores indicate greater chronic stress severity
Mental toughness | Within the 6 months after intervention randomization
  Sports Mental Toughness Questionnaire (SMTQ); Scale ranges from 5-25; Higher scores indicate higher confidence & constancy
History of suicidal ideation, plan, & attempt | Within the 6 months after intervention randomization
  Columbia-Suicide Severity Rating Scale (C-SSRS) Full scale Baseline/Screening; Scale ranges from 0-1 0=No; 1=Yes
Positive social networks | Within the 6 months after intervention randomization
  Supportive & Negative Social Interaction Scale (SIS); Scale ranges from 0-8; Higher scores indicate more positive/negative social support
Negative social networks | Within the 6 months after intervention randomization
  Supportive & Negative Social Interaction Scale (SIS); Scale ranges from 0-8; Higher scores indicate more positive/negative social support
Mattering/belonging | Within the 6 months after intervention randomization
  General Mattering Scale; Scale ranges from 0-20; Higher scores indicate higher perceived mattering to others
Loneliness | Within the 6 months after intervention randomization
  3-Item Loneliness Screener; Scale ranges from 0-16; Higher scores indicate more frequency-severity of loneliness
Adverse childhood events & trauma | Within the 6 months after intervention randomization
  Childhood Trauma Questionnaire - Short Form (CTQ-SF) ; Scale ranges from 0-44; Higher scores indicate more childhood maltreatment
Conscientiousness | Within the 6 months after intervention randomization
  Big Five Inventory (BFI)16 & Personality Inventory for DSM-5 Brief Form (PID-5-BF); Scale ranges from 0-8; Higher scores indicate lower of each adaptive trait
Mastery | Within the 6 months after intervention randomization
  Pearlin & Schooler's Psychological Coping Resources Measure; Scale ranges from 0-8; Higher scores indicate lower of each adaptive trait
Openness | Within the 6 months after intervention randomization
  120-item International Personality Item Pool (IPIP); Scale ranges from 0-4; Higher scores indicate lower of each adaptive trait
Problem-solving ability | Within the 6 months after intervention randomization
  Social Problem Solving Inventory-Revised (SPSI-R); Scale ranges from 0-8; Higher scores indicate lower of each adaptive trait
Psychological well-being | Within the 6 months after intervention randomization
  Flourishing Scale; Scale ranges from 0-12; Higher scores indicate lower of each adaptive trait
Resilience | Within the 6 months after intervention randomization
  Army STARRS Resilience Scale; Scale ranges from 0-16; Higher scores indicate lower of each adaptive trait
Self-esteem | Within the 6 months after intervention randomization
  Rosenberg Self-Esteem Scale; Scale ranges from 0-8; Higher scores indicate lower of each adaptive trait
Anxious, Cyclothymic, Depressive, & Hyperthymic temperament | Within the 6 months after intervention randomization
  Revised NEO Personality Inventory (NEO-PI-R) & the Temperament Evaluation of Memphis, Pisa, Paris & San Diego-autoquestionnaire version (TEMPS-A); Scale ranges from 0-8 for each temperament; Higher scores indicate higher of each maladaptive trait
Borderline personality | Within the 6 months after intervention randomization
  McLean Screening Instrument for Borderline Personality Disorder; Scale ranges from 0-16; Higher scores indicate higher of each maladaptive trait
Anger-hostility | Within the 6 months after intervention randomization
  Big Five Inventory (BFI)16 & Personality Inventory for DSM-5 Brief Form (PID-5-BF); Scale ranges from 0-8; Higher scores indicate higher of each maladaptive trait
Impulsivity/negative urgency | Within the 6 months after intervention randomization
  Impulsive Behavior Scale - Short Form (SUPPS-P); Scale ranges from 0-8; Higher scores indicate higher of each maladaptive trait
Introversion | Within the 6 months after intervention randomization
  Eysenck Personality Questionnaire - Brief Version (EPQ-BV)28 & Revised NEO Personality Inventory (NEO-PI-R); Scale ranges from 0-8; Higher scores indicate higher of each maladaptive trait
Fearlessness about death | Within the 6 months after intervention randomization
  Acquired Capability for Suicide Scale; Scale ranges from 0-4; Higher scores indicate higher of each maladaptive trait
Self-conscious | Within the 6 months after intervention randomization
  Widiger Five-Factor Rating Form - Revised31 & NEO Five-Factor Inventory (NEO-FFI); Scale ranges from 0-8; Higher scores indicate higher of each maladaptive trait
Vulnerability | Within the 6 months after intervention randomization
  NEO Five-Factor Inventory (NEO-FFI); Scale ranges from 0-4; Higher scores indicate higher of each maladaptive trait
Frequency of risky behaviors | Within the 6 months after intervention randomization
  Unit Risk Inventory (URI); Scale ranges from 0-1; 0=Never; 1=At least less than once a month

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Nassif, PhD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Fort Hood Installation Reception Center, Fort Hood, Texas, United States

IPD SHARING:
Plan to Share IPD: No